CLINICAL TRIAL: NCT02366286
Title: Hepatitis B and Hepatitis C as Risk Factors for Hepatocellular Carcinoma in African and Asian Immigrants: Role of Viral Genetics and the Immune Response
Brief Title: Hepatitis B and Hepatitis C as Risk Factors for Hepatocellular Carcinoma in African and Asian Immigrants
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Gargar Clinic (Other); Axis Medical Center (Unknown)
Responsible Party: Sponsor
Other Study IDs: 09-001670; IN-US-174-0230 (Other Grant/Funding Number: Gilead)
Record Dates: First submitted 2014-10-08; First posted 2015-02-19 (Estimated); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Hepatitis B; Hepatitis C; Carcinoma, Hepatocellular
MeSH Terms: conditions — Hepatitis B; Hepatitis C; Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A blood draw of 45 ml. will be taken for serum, plasma and buffy coat
Oversight: Data Monitoring Committee: No

SUMMARY:
The prevalence of hepatitis B virus (HBV) and hepatitis C virus (HCV) in the United States (US) is relatively low. However, immigrant populations in the US from Asia and sub-Saharan Africa have substantially higher prevalence than the general population and are consequently at a significant risk for hepatocellular carcinoma (HCC). Indeed, the age-adjusted incidence rates for HCC in the US have tripled from 1975 to 2005. As the population demographics have changed, the 2000 US census estimated the number of Somalis in Minnesota at 25,000 but current estimates put the number at around 50,000 due to primary refugee arrivals as well as secondary immigration from other states. There is no available data for Somali immigrants in the US on HBV and HCV prevalence, HBV and HCV genotypes/subgenotypes, and genetic and immunologic risk factors predisposing Somalis to HBV and HCV and the subsequent development of HCC. Therefore. this study will fill these gaps in the Somali population to understand the relative importance of HBV and HCV infections in causation of HCC.

Besides Somalis, Minnesota is also home to large other African immigrant communities. According to the Minnesota Department of Health (MDH), in 2013, the highest rates of chronic HBV cases where reported among Asian or Pacific Islanders (3,638 cases per 100,000 persons) followed by Black or African Americans (2,078 cases per 100,000 persons). Additionally, Minnesota receives a large number of new refugee's resettlement. It is important to improve the identification of chronic HBV and HCV infections among Somali refugees and immigrants in Minnesota through well-designed community-wide screening efforts. Since we know that African immigration to Minnesota is the third highest in the US, this unique population might be a contributing factor to the increased burden of hepatitis and liver cancer complications in the state of Minnesota. Findings from HBV and HCV screening among Somalis suggest that other immigrant African populations from high viral hepatitis endemic regions, such Ethiopia, Liberia, and Kenya, are also at substantial risk of HBV, HCV and HCC. Unfortunately, very little research has been conducted in the US on the burden of hepatitis and liver cancer in African Immigrants from areas of high endemicity of hepatitis B and hepatitis C. Therefore, the goal of is to identify HBV and HCV and the role viral genetics and immune response among African immigrant communities from Kenya, Liberia, and Ethiopia.

DETAILED DESCRIPTION:
Specific Aim 1: We will determine whether exposures to HBV and HCV infections in African (Somalis, Kenyans, Liberians, and Ethiopians) and Southeast Asian (Hmong, Vietnamese, Laotian, and Cambodian) are associated with a single HBV/HCV genotype or few specific subtypes. In the following Sub-Aims we will:

* confirm the viral status of study subjects using serological and DNA tests including HBsAg, HBcAb, anti-HCV, HBV DNA and HCV RNA.
* perform nucleic acid testing to identify the HBV and HCV genotypes/sub-genotypes for each patient
* examine the presence of either common or unique HBV and HCV viral mutations

Specific Aim 2: We will determine whether African (Somalis, Kenyans, Liberians, and Ethiopians) and Southeast Asian (Hmong, Vietnamese, Laotian, and Cambodian) exposed to HBV or HCV have unique TLR or Treg immune signatures as compared to control subjects free from both HBV and HCV infections. In the following Sub-Aims we will:

* measure the expression levels of toll-like receptors (in monocytes) of the host innate immune response to assess whether the expression of TLR differs between those exposed to HBV vs HCV
* measure the circulating Tregs of the host adaptive immune response to determine whether the abundance of Treg differs between those exposed to HBV vs HCV Specific Aim 3: To determine whether genetic variation of IL28B (assessed by single nucleotide polymorphisms, rs12979860 and others) is associated with HCV treatment outcome in Somalis.
* We will perform SNP analysis of IL28B in lymphocyte DNA in 60 HCV cases, 60 HBV and HCV cases and 60 healthy controls (this group and additional 60 HBV cases alone will provide baseline SNP frequencies in the Somali population), all the 240 subjects of the study will be tested for this SNP
* We will measure treatment outcome using virological response by comparing pre-treatment viral load and post-treatment viral load in HCV case

Aim 4: To recruit a cohort of African (Somalis, Kenyans, Liberians, and Ethiopians) and Southeast Asian (Hmong, Vietnamese, Laotian, and Cambodian)immigrants for screening for chronic HBV infection and education on prevention and treatment of hepatitis B. We will specifically:

* Establish a community-based program to recruit African and Southeast Asian individuals in Minnesota for screening for hepatitis B and hepatitis C
* Establish partnerships with African and Southeast Asian community organizations and physicians to enhance screening and education about prevention and treatment of hepatitis B, hepatitis C and its sequelae, including HCC.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* African descent
* Southeast Asian descent

Exclusion Criteria:

* 17 years or younger

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: African and Southeast Asian immigrant and refugees
Sampling Method: Non-Probability Sample
Enrollment: 892 (Actual)
Dates: Start 2010-11 (Actual); Primary Completion 2017-09-11 (Actual); Study Completion 2017-10-05 (Actual)

PRIMARY OUTCOMES:
Number of subjects who test positive for markers of Hepatitis B Virus infection (HBsAg, HBcAb, HBsAb) | 2 Years
Number of subjects who test positive for markers of Hepatitis C Virus infection (anti-HCV infection) | 2 years
Rate of HBV vaccination in subjects with negative HBV serology | 2 Years

SECONDARY OUTCOMES:
Incidence of HCC over the period of the study | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Lewis R. Roberts, MB ChB, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials